CLINICAL TRIAL: NCT01102855
Title: Confocal Laser Endomicroscopy in Patients With Crohn´s Disease
Brief Title: Endomicroscopy and Crohn´s Disease
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Markus F. Neurath, M.D., Ph.D., University of Erlangen-Nuremberg
Other Study IDs: HN-0002
Record Dates: First submitted 2010-04-12; First posted 2010-04-13 (Estimated); Last update posted 2011-08-11 (Estimated); Status verified 2011-08

CONDITIONS: Crohn´s Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Purpose:

The main objective of this study is to determine endomicroscopic features of Crohn´s disease.

Background:

Crohn´s disease is an inflammatory disease of the intestines that may affect any part of the gastrointestinal tract from anus to mouth, causing a wide variety of symptoms. Diagnosis is based on several histologic features including transmural pattern of inflammation, crypt abscesses and granulomas. Confocal laser endomicroscopy (CLE) is rapidly emerging as a valuable tool for gastrointestinal endoscopic imaging, enabling the endoscopist to obtain an "optical biopsy" of the gastrointestinal mucosa during the endoscopic procedure.

Scope:

In patients with Crohn´s disease.

DETAILED DESCRIPTION:
Methods:

Patients underwent colonoscopy for the evaluation of Crohn´s disease. During the endoscopic procedure CLE will be performed.

Procedure:

The patient underwent colonoscopy. During the procedure the patient will receive intravenous fluorescein or topical mucosal staining with acriflavin or cresyl violet, followed by in-vivo CLE of the tissue. Confocal images are digitally saved and analyzed afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age 18-85 years
* Ability of subjects to understand character and individual consequences of clinical trial
* Subjects undergoing colonoscopy

Exclusion Criteria:

* Inability to provide written informed consent
* Severe Coagulopathy (Prothrombin time < 50% of control, Partial thromboplastin time > 50 s)
* Impaired renal function (Creatinine > 1.2 mg/dl)
* Pregnancy or breast feeding
* Active gastrointestinal bleeding
* Known allergy to fluorescein, acriflavin or cresyl violet
* Residing in institutions (e.g. prison)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Crohn´s disease.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2009-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
To determine endomicroscopic features of Crohn´s disease. | October 2009 until May 2010

SECONDARY OUTCOMES:
Comparison of CLE findings with conventional histology. | October 2009 until May 2010

CONTACTS AND LOCATIONS:
Overall Officials: Markus F. Neurath, Study Director — University of Erlangen-Nürnberg
Locations (1):
- Department of Medicine I, University of Erlangen-Nuremberg, Erlangen, Germany

REFERENCES:
- [Derived] Neumann H, Vieth M, Atreya R, Grauer M, Siebler J, Bernatik T, Neurath MF, Mudter J. Assessment of Crohn's disease activity by confocal laser endomicroscopy. Inflamm Bowel Dis. 2012 Dec;18(12):2261-9. doi: 10.1002/ibd.22907. Epub 2012 Feb 16. PMID 22344873